CLINICAL TRIAL: NCT03212859
Title: Coach2Move: Sustainable in Daily Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 104612
Record Dates: First submitted 2017-06-28; First posted 2017-07-11 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Sedentary Lifestyle; Physical Activity; Frail Elderly Syndrome
Keywords: older adults; physiotherapy; physical activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: stepped wedge cluster randomised trial and mixed methods process analysis
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coach2Move Intervention Group (Experimental): Coach2Move Intervention Group
  Interventions: Behavioral: Coach2Move
- Usual Care (Active Comparator): Usual care physiotherapy among older adults
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Coach2Move — Coach2Move is a multicomponent physiotherapeutic approach in addition to usual care physiotherapy consisting of:
  * Extensive intake during which not only impairments and disabilities, but wishes, barriers and facilitators considering physical functioning are profoundly examined.
  * Motivational interviewing is used to find and deal with barriers for becoming physically active and shared-decision making in goal setting.
  * The approach is patient focused (tailor made) and goal-oriented: the physiotherapist coaches the patient and the environment in reaching and maintaining their own goals.
  * In consultation with the patient, a stratified intervention is chosen by picking the best fitting option out of three patient-tailored intervention profiles with a predefined number of intervention sessions.
  Arms: Coach2Move Intervention Group
Behavioral: Usual Care — Usual care physiotherapy among older adults:
  * Intake of 30 minutes consisting of examining medical history, physical functioning and functional exercises to assess the demand for care.
  * Use of treatment modalities to enhance physical functioning (strength, mobility, coordination, balance etc.)
  * Consultation and advisory role in relation to the functional status of geriatric patients and his/her relations.
  * Collaborate with other disciplines in a multidisciplinary context.
  Arms: Usual Care

SUMMARY:
Implementation of a previously shown (cost-)effective physical therapeutic treatment strategy for community-dwelling older adults.

DETAILED DESCRIPTION:
In a previous trial, researchers demonstrated that the Coach2Move approach is superior to regular physiotherapy in terms of increasing physical activity, reducing frailty, improving quality of life and reducing healthcare costs. In short, in less physiotherapeutic sessions, better outcomes were realized.

Despite these promising findings, the research group still has questions regarding the generalisability of these findings. The reservations towards the generalisability of the approach are caused by the following:

1. A modest (n=130), yet somewhat selective study sample was included: nearly half of the eligible individuals declined randomisation and thereby participation. An understanding is needed how this group of eligible non volunteers respond to Coach2Move. Therefore, a study design that avoids randomisation at the patient level will be used.
2. The Coach2Move approach significantly increased the level of moderate physical activity among the treatment group and reduced levels of frailty significantly after 6 months, but the clinical importance of these findings is still unclear. Thus, a replication of the effects in the light of physical functioning is needed in a larger more variable study population and with a longer follow-up.

In addition, the results from the earlier carried out RCT concerning the cost-effectiveness of Coach2Move have to be replicated on a larger scale.

For the reasons mentioned above, it is important to further implement Coach2Move and study its effect, costs, and feasibility in current practice. A stepped wedge cluster randomised trial design is chosen because in the opinion of the researchers, the implementation strategy will do more good than harm (making a parallel design, in which certain practices do not receive the intervention or to withdraw the intervention as would occur in a cross-over design, is unethical) and it furthermore minimizes contamination.

The objective of this study is to assess the cost-effectiveness of the implementation of a patient and context focused tailored coaching intervention (Coach2Move) in the daily physiotherapy practice for older adults with mobility problems compared to usual physiotherapy. The hypothesis is that Coach2Move leads to better physical outcomes and lower costs than usual care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Community-dwelling
* mobility related problems or problems related to activities of daily living
* sedentary lifestyle or are at risk of losing an active lifestyle

Exclusion Criteria:

* Patients who are not ambulatory after treatment and/or are in palliative phase.
* Patients who are indicated to become institutionalised in the near future.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 292 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Self-reported Physical Activity | 27 months
  The primary outcome of the study is physical activity measured by the LAPAQ questionnaire, subscale moderate activity. This subscale of the LAPAQ is a comprehensive questionnaire on diverse (physical) activities of daily living with moderate intensity including walking, riding a bicycle etc. and is specifically designed to assess habitual physical activity of the elderly.
Functional Mobility | 27 months
  The key secondary outcome is functional mobility as measured by the Timed Up and Go test.

SECONDARY OUTCOMES:
Functional Status | 12 months
  The Patient Specific Complaints Scale is used to measure the functional status of a patient. The patients select 3-5 most important mobility problems in daily life and are the most important goals to improve. The degree of hinder is scored by the patient on a 10-point numeric scale.
Cost effectiveness | 27 months
  The direct costs of regular physiotherapy and Coach2Move will be determined on a per patient basis. On patient level, volumes of care will be measured prospectively using medical records and cost questionnaires.
  Next will be determining the cost prices for each volume of consumption in order to use these for the volumes registered for each participating patient.
  Both outcome measures will be aggregated to one reported value (cost per volume x volumes used). A comparison in costs will be made between the Coach2Move and usual care groups.
Patient Satisfaction | 27 months
  The Global Perceived Satisfaction and Effect score is used to measure the patients' satisfaction about the intervention and the perceived effect on a 7-point Likert scale ranging from very unsatisfied to very much satisfied and very much deterioration to very much improvement, respectively.
Level of Frailty | 27 months
  To measure the level of frailty and participation, the Evaluative Frailty Index is used. This questionnaire consists of 50 items on deficits in health (symptoms, signs and disabilities) in multiple domains (physical, psychological, social and general health status).

OTHER OUTCOMES:
Implementability | 27 months
  group interviews with PT's and PTG's within each practice will inform us about views and experiences of facilitators and barriers in delivering the Coach2Move interventions and views on which elements on the Coach2Move were effective and which were not, and if the education, peer assessment, EPD, and measurement procedures were viewed as helpful or unhelpful in supporting them to realize behavioural change strategies including needs assessment, problem analysis, shared decisions on SMARTI goals, and monitoring feedback
Budget Impact | 27 months
  lts purpose is to estimate the financial consequences of adoption and diffusion of standard use of the Coach2Move approach in the Netherlands. Several scenarios will be evaluated. The aim is to assess these consequences in the medium-long term from the various budget holders' perspectives 1) wider societal perspective; 2) the more narrow perspective of the public purse; 3) the perspective of the health insurers; 4) the perspective of the health care provider.
  The Budget Impact Analysis will be assessed through modelling and analysed in a probabilistic way.
  Deterministic uncertainty concerning the analysis' input such as the perspective, pricing parameters, time horizon, uptake, etc. will be dealt with by generating the budget impact as a series of scenario analyses covering a relevant range of costs.

CONTACTS AND LOCATIONS:
Overall Officials: Ward Heij, MSc, Principal Investigator — Radboud University Medical Center
Locations (1):
- Ward Heij, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heij W, Sweerts L, Staal JB, Teerenstra S, Adang E, van der Wees PJ, Nijhuis-van der Sanden MWG, Hoogeboom TJ. Implementing a Personalized Physical Therapy Approach (Coach2Move) Is Effective in Increasing Physical Activity and Improving Functional Mobility in Older Adults: A Cluster-Randomized, Stepped Wedge Trial. Phys Ther. 2022 Dec 6;102(12):pzac138. doi: 10.1093/ptj/pzac138. PMID 36200397
- [Derived] Heij W, Teerenstra S, Sweerts L, Staal JB, Nijhuis-van der Sanden MWG, Hoogeboom TJ. Implementation of a Cost-Effective Physical Therapy Approach (Coach2Move) to Improve Physical Activity in Community-Dwelling Older Adults With Mobility Problems: Protocol for a Cluster-Randomized, Stepped Wedge Trial. Phys Ther. 2020 Apr 17;100(4):653-661. doi: 10.1093/ptj/pzz183. PMID 31846501
- See also: Previous Trial — https://www.ncbi.nlm.nih.gov/pubmed/27239405
- See also: Previous Trial — https://www.ncbi.nlm.nih.gov/pubmed/25621385

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT03212859/Prot_SAP_000.pdf